CLINICAL TRIAL: NCT03107598
Title: Colloid Preload Versus Crystalloid Co-load in Cesarean Section Under Spinal Anesthesia Randomized Controlled Trial
Brief Title: Colloid Preload Versus Crystalloid Co-load in Cesarean Section Under Spinal Anesthesia
Acronym: CPvsCC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Mahdia (Other)
Responsible Party: Principal Investigator, Majdoub Ali MD, head of anesthesia department clinical professor, University Hospital, Mahdia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LCS
Record Dates: First submitted 2016-12-30; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Hypotension
Keywords: spinal anesthesia; neonatal outcome; Caesarean Section
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- colloid preload (Experimental): Group CoP: group with colloid preload The preload group received rapid infusion of 15ml/kg of 6% hydroxyethyl starch (6% HES) administered by gravity at a wide-open rate over a period of 15-30min before induction of spinal anesthesia.
  Interventions: Drug: colloid preload
- crystalloid coload (Placebo Comparator): Group CrC: group with crystalloid coload The coload group received a sodium chloride 0.9% perfusion as rapidly as possible starting at the time of intrathecal injection for spinal anesthesia.
  Interventions: Drug: colloid preload

INTERVENTIONS:
Drug: colloid preload — coparaison between colloid and crystalloide loading in spinal anesthesia for cesarean section
  Other Names: crystalloid coload

SUMMARY:
Comparison between colloid preload and crystalloid co-load in cesarean section under spinal anesthesia.

1. The primary outcome was the incidence of hypotension
2. Secondary outcomes included the incidence of severe hypotension, total ephedrine dose, nausea and vomiting and neonatal outcome assessed by Apgar scores and umbilical artery blood gas analysis

DETAILED DESCRIPTION:
It's a prospective randomized study, during 7 months between march and September 2016, carry on department of anesthesia and intensive care and department of obstetrics and gynecology, at Taher Sfar Mahdia University Hospital. investigators included participants:

* Aged between 18 and 40 years' old
* American Society of Anesthesiologists physical status I or II (ASA)
* Full-term singleton pregnancy
* scheduled for elective cesarean section under spinal anesthesia

Parturients were excluded if :

* participants younger than 18 or older than 40 years
* cardiovascular, cerebrovascular or renal disease
* multiple gestations
* polyhydramnios or known fetal abnormalities
* allergy to local anesthetics or opioids
* emergency Cesarean section or parturient that have failed vaginal delivery with epidural analgesia
* contraindications for performing spinal anesthesia in this study no premedication was given. Patients entered the operating room and lay supine with 15° of left lateral tilt on the operating table.

Standard monitors of electrocardiography, pulse oximetry (Spo2), and noninvasive blood pressure were applied on the right arm.

Baseline systolic and diastolic blood pressure (SBP, DPB) and heart rates (HR) were recorded. An 18 or 16-gauge intravenous cannula was inserted in a large forearm vein.Patients were randomly assigned into two groups: colloid preload (CoP), and crystalloid co-load (CrC).Group CoP: group with colloid preload The preload group received rapid infusion of 15ml/kg of 6% hydroxyethyl starch (6% HES, voluven) administered by gravity at a wide-open rate over a period of 15-30min before induction of spinal anesthesia.Group CrC: group with crystalloid coload received a sodium chloride 0.9% perfusion as rapidly as possible starting at the time of intrathecal injection.

Spinal anesthesia was performed in the sitting position with a 27- or 25-gauge spinal needle at the L3-4 or L2-3 interspace using hyperbaric bupivacaine 10 mg (0.5% hyperbaric bupivacaine 2 mL), sufentanyl 2.5 µg (0.5 ml) and 100µg morphine (1ml). All patients received the same dose regardless of height or weight. After completing the anesthetic procedure, patients were immediately repositioned to supine with a 15°-30° left lateral tilt. The highest sensory block was checked and confirmed at the level of T3-T5 determined with loss-to-pinprick method bilaterally at 5 minutes and 10 minutes after spinal drug administration. Motor block was measured with modified Bromage scale (0, no block; 1, inability to raise extended leg;2, inability to flex knee; 3, inability to flex ankle and foot).

Oxygen was routinely given: 5 l/min was administrated via a clear facemask. After umbilical cord clamping, prophylactic antibiotic treatment was administrated intravenously whether 2g of cefazolin or 600mg of clindamycin if the parturient was allergic to penicillin.After delivery of the baby, 10 UI of oxytocin was intravenously given, and 15 UI was titrated following lactate ringer's solution.

Hypotension was defined as a 20% reduction of systolic blood pressure from baseline .Severe hypotension defined as SBP < 80 mmhg.

It was treated with an intravenous ephedrine bolus:

* 70% ≤ SBP < 80% from baseline value: ephedrine 6mg
* SBP < 70% from baseline value: ephedrine 9mg
* SBP < 60% from baseline value: ephedrine 12mg Vasopressor treatment was repeated every 2 minutes if hypotension persisted or recurred.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40 years' old
* American Society of Anesthesiologists physical status I or II (ASA)
* Full-term singleton pregnancy
* scheduled for elective cesarean section under spinal anesthesia

Exclusion Criteria:

* cardiovascular, cerebrovascular or renal disease
* multiple gestations
* polyhydramnios or known fetal abnormalities
* allergy to local anesthetics or opioids
* emergency Cesarean section or parturient that have failed vaginal delivery with epidural analgesia
* contraindications for performing spinal anesthesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the incidence of hypotension | 2 hours
  hypotension defined by decreasing of arterial blood pressure under 20% of base line

SECONDARY OUTCOMES:
incidence of severe hypotension | 2 hours
  severe hypotension is defined by decreasing of systolic arterial blood pressure below 80 mmHg
total ephedrine dose | 2 hours
nausea and vomiting | 2 hours
  number of nausea and vomiting episode
neonatal outcome | 2 hours
  umbilical arterial blood gas and APGAR scors at 1 and 5 minutes

IPD SHARING:
Plan to Share IPD: No